CLINICAL TRIAL: NCT03360448
Title: Randomized, Phase 3, Placebo-Controlled Double-Blind, Multicenter Trial of a One Time Intracoronary Administration of Ad5.hAC6 Gene Transfer for Patients With Reduced Left Ventricular Heart Failure
Brief Title: AC6 Gene Transfer in Patients With Reduced Left Ventricular Ejection Fraction Heart Failure
Acronym: FLOURISH
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Clinical development plans and strategy for RT-100 being re-evaluated
Sponsor: Renova Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT-01-HF-REF
Record Dates: First submitted 2017-11-13; First posted 2017-12-04 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure
Keywords: Gene Transfer
MeSH Terms: conditions — Heart Failure | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Ad5.hAC6: Intracoronary delivery of adenovirus encoding human adenylyl cyclase type 6
  Interventions: Drug: Ad5.hAC6
- Placebo Comparator (Placebo Comparator): Placebo: Intracoronary delivery of formulation buffer ( 3% sucrose)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ad5.hAC6 — 1:1 randomization (Ad5.hAC6 : placebo) - intracoronary delivery
  Other Names: RT-100
  Arms: Experimental
Drug: Placebo — 1:1 randomization (Ad5.hAC6 : placebo) - intracoronary delivery
  Other Names: 3% sucrose
  Arms: Placebo Comparator

SUMMARY:
To determine the safety and efficacy of an intracoronary injection of adenovirus 5 encoding human adenylyl cyclase 6 (RT-100) in patients with heart failure with reduced left ventricular ejection fraction (HFrEF) in a Phase 3 clinical trial.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded Phase 3 clinical trial using a one-time intracoronary injection of Ad5.hAC6 (or placebo) to determine safety and efficacy in patients with documented HFrEF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years, inclusive, with history of heart failure (HF).
2. Current HF symptoms with NYHA Functional Classification Class II to IV (inclusive) at Screening (Visit 1).
3. Currently receiving optimally tolerated standard of care HF medical therapy as defined by the American Heart Association (AHA)/American College of Cardiology (ACC) Heart Failure guidelines and Focused Update along with an angiotensin converting enzyme inhibitor (ACEi)/angiotensin II receptor blockers (ARB), diuretics and sacubitril/valsartan for 4 weeks or longer, without change in drug therapy or dosage regimen, prior to Visit 1 (and continued same HF therapy through Visit 2).
4. Left Ventricular Ejection Fraction (LVEF) ≥ 10 to ≤ 35% as determined by Screening echocardiogram (ECHO).
5. NT pro BNP ≥ 400 pg/mL.
6. If subject has had coronary artery bypass surgery, then at least one conduit must be patent and therefore be amendable for test article.
7. Women of child bearing capacity must have a negative pregnancy test before 2 days of test article administration and must not be currently breastfeeding or nursing, and female and male patients must be willing to use birth control for 12 weeks after test article administration if the female partner is of child bearing capacity. Acceptable methods of effective birth control include total sexual abstinence; a condom with spermicide (men) in combination with barrier methods (diaphragm, cervical cap or cervical sponge); hormonal birth control (oral or injectable contraceptives); intrauterine devices; or surgical sterilization (vasectomy and testing that shows there is no sperm in the semen for men and bilateral tubal ligation +/- oophorectomy for women).
8. Willing to provide informed consent consistent with International Conference on Harmonisation Good Clinical Practices.

Exclusion Criteria:

1. Use of intravenous (IV) vasodilatory or inotropic therapy within 24 hours prior to Visit 2.
2. Unstable angina within 3 months of Visit 1.
3. Coronary revascularization planned or predicted within 6 months prior to Visit 1.
4. Subjects who are candidates for revascularization are not considered appropriate for this trial; therefore, if a subject has Ischemia of viable myocardium > 15% and is a candidate for revascularization, this subject would not be eligible to participate in this trial.
5. Myocardial infarction within 6 months prior to Screening (Visit 1). Myocardial infarction is defined by documented evidence of a rise and/or fall of cardiac biomarker values (preferably cardiac troponin) with at least one value above the 99th percentile upper reference limit, and either ischemic symptoms, electrocardiogram changes, imaging evidence of loss of viable myocardium or new regional wall motion abnormality, or identification of an intracoronary thrombus by coronary angiography.
6. Thrombocytopenia (< 100,000 platelets/µL) or bleeding diathesis.
7. Stroke or transient ischemic attack within 6 months prior to Screening (Visit 1).
8. Use of sodium-glucose co-transporter 2 inhibitors used to treat type 2 diabetes mellitus.
9. Cardiac:

   1. Biopsy documenting reversible cause of cardiomyopathy within 6 months of Visit 1 (Screening) if available as part of patient's prior cardiac history.
   2. Acute cardiac decompensation.
   3. If coronary angiogram within 6 months, with a presence of untreated severe three vessel coronary disease or unprotected left main coronary artery disease or coronary anatomy unsuitable for study procedure (eg, arterial tortuosity, etc) prior to Randomization (Visit 2).
   4. Use of IV diuretics within 12 hours of Randomization (Visit 2).
   5. Hemodynamically significant untreated valvular heart disease based on the AHA/ACC Valvular Heart Disease Guidelines.
   6. Current evidence of restrictive, peripartum, viral, infectious, infiltrative, or inflammatory cardiomyopathy.
   7. Significant pericardial effusion at Screening (Visit 1) or at the time of test article administration.
   8. Current untreated ventricular arrhythmias.
   9. Currently awaiting planned heart transplantation or ventricular assist device.
   10. Congenital heart disease (other than small or hemodynamically non significant ventricular septal defect or atrial septal defect).
   11. Device therapy as noted below:

   i. Cardiac resynchronization therapy (CRT), or CRT-D/P, is not allowed within 6 months of implantation.

   ii. Implantable Cardioverter Defibrillator or pacemaker implantation is not allowed if implanted < 30 days prior to Screening (Visit 1).

   iii. CardioMems device is not allowed.

   l. Systolic blood pressure ≥ 160 mm Hg or < 90 mm Hg at Visit 1 or 2.

   m. Diastolic blood pressure ≥ 95 mm Hg at Visit 1 or 2.
10. 6 Minute Walk Test (6MWT):

    1. Inability to perform the 6MWT for reasons unrelated to heart failure (eg, physical limitations, peripheral vascular disease).
    2. Distance walked in 6MWT (6MWD) < 100 m
11. Pulmonary:

    1. Pulmonary disease requiring oxygen therapy;
    2. Severe chronic obstructive pulmonary disease; restrictive lung disease.
12. Upper respiratory infection within 4 weeks of Screening (Visit 1).
13. History of organ transplant.
14. Viral syndrome with fever ≥101° Fahrenheit (patient may be reconsidered for enrollment 4 weeks following resolution of viral syndrome).
15. History of human immunodeficiency virus or acquired immunodeficiency syndrome, history of hepatitis C virus, or immunosuppressed by medicines (corticosteroids, methotrexate, cyclophosphamide, cyclosporine).
16. Presence of eGFR ≤ 30 mL/min/1.73 m2 using the Cockcroft Gault equation.
17. Patients with life expectancy < 1 year.
18. Documented Child Pugh B or C hepatic disease.
19. Body Mass Index ≥ 40 kg/m2.
20. Participation in any other clinical trial or registry within 30 days prior to Randomization (Visit 2).
21. Hemoglobin ≤ 10 gm/dL.
22. Prior history of malignancy.
23. Prior history of gene transfer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Hospitalizations | Baseline to 12 months
  Reduce the event rate of all (first and repeat) heart failure hospitalizations

SECONDARY OUTCOMES:
Cardiovascular (CV) Death | Baseline to 12 months
  Reduce the event rate of cardiovascular (CV) death
All Cause Death | Baseline to 12 months
  Reduce the event rate of death (regardless of cause)
New York Heart Association (NYHA) Functional Classification | Baseline to 12 months
  Improve NYHA functional classification
All Heart Failure (HF) Events | Baseline to 12 months
  Reduce the event rate of all heart failure (HF) events

OTHER OUTCOMES:
Echocardiographic Parameters | Baseline to 12 months
  Improve echocardiographic parameters of left ventricular systolic and diastolic functions.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to 12 months
  Improve clinical summary score for heart failure (HF) symptoms and physical limitations as assessed by KCCQ. Scores will be calculated according to the guidance provided by CV Outcomes Inc.
Six Minute Walk Distance | Baseline to 12 months
  Improve the six-minute walk distance (6MWD) using the standard according to the American Thoracic Society March 2002 Guidelines using a 100 foot hallway or corridor
Borg Dyspena Score | Baseline to 12 months
  Improve the Borg dyspnea score. The Borg Scale will be used (0-10, 0 = nothing at all, 10 = very, very severe)
NT-proBNP | Baseline to 3 and 12 months
  Improve N-terminal pro brain natriuretic peptide (NT-proBNP)

IPD SHARING:
Plan to Share IPD: Undecided
Blinded study - de-identified participant data to become available after completion of study.

REFERENCES:
- [Background] Hammond HK, Penny WF, Traverse JH, Henry TD, Watkins MW, Yancy CW, Sweis RN, Adler ED, Patel AN, Murray DR, Ross RS, Bhargava V, Maisel A, Barnard DD, Lai NC, Dalton ND, Lee ML, Narayan SM, Blanchard DG, Gao MH. Intracoronary Gene Transfer of Adenylyl Cyclase 6 in Patients With Heart Failure: A Randomized Clinical Trial. JAMA Cardiol. 2016 May 1;1(2):163-71. doi: 10.1001/jamacardio.2016.0008. PMID 27437887